The Use of Delta-Wave Hypnoanalgesia as a Non-Pharmacological Adjunct to Reduce Perioperative Anxiety During Cataract Surgery: A Prospective Randomized Single-Blind Study

## Statistical Analysis:

Distribution normality for numerical data was tested by the Kolmogorov–Smirnov test. Descriptive study was conducted by calculating the mean of diverse studied variables. Continuous variables were compared using Student's t-tests, and categorical variables using chi-square tests. We performed all statistical analyses with SPSS statistical software version 22.0 (SPSS Inc., Chicago, IL, USA) and Excel Microsoft Office. A p-value <0.05 was considered statistically significant.